CLINICAL TRIAL: NCT04557592
Title: Comparisons of gaIt aNalyses pERformance Between the Gaitrite walkwaYs
Acronym: CINERGY
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020/110
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Gait Apraxia; Alzheimer Disease; Impaired Cognition
MeSH Terms: conditions — Gait Apraxia; Alzheimer Disease; Cognition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The GAITRite® system is an instrumented with resistive pressure sensors gait analyzer. It was first validate in 2001 against paper-and-pencil (intraclass correlation coefficient [ICC] > 95%) for spatial measures and against video-based (ICC > 93%) for temporal measures, and was thus a reliable tools to measure step lengths and times in both walkway center and left-of-center measurements. It was considered as one of the gold standards in gait analyses. This gait analyze system may distinguish prospectively faller and non-faller older adults, but it can detect spatial, temporal, and spatiotemporal measures of gait and greater variability of gait parameters which were associated with and predictive of both global- and domain-specific cognitive decline. Moreover, spatiotemporal gait parameters analyzed using GAITRite® were more disturbed in the advanced stages of dementia, and more affected in the non-AD dementia than in AD suggesting that quantitative gait parameters could be used as a surrogate marker for improving the diagnosis of dementia.

Nevertheless, GAITRite® is not a unique system and it comprises different walkways. One of these technologies was a roll-up system (platinum plus classic, RE, Basic and Safari), and the other was a system composed by a changeable association of plates (CIRFACE). In order to ensure a good comparability between studies using these different walkways, it appears important to compare the performances of these walkways in gait analysis. Thus, the main aim of this study was to compare the performances in gait analyze between the GAITRite® platinum plus classic and the GAITRite® CIRFACE among older adults. Secondary aims were to compare these parameters among patients with cognitive complaint, minor or major neurocognitive disorder (NCD) related to Alzheimer disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 75 years
* Gait analysis performed with the two walkways superimposed during a consultation or day hospitalization

Exclusion Criteria:

* Opposition to the use of the information collected for research purposes

Min Age: 74 Years | Sex: All
Age Groups: Older Adult
Study Population: All consecutive patients meeting the eligibility criteria over the study period.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Change in spatiotemporal gait, and in particular in the variability of stride time between the two devices | baseline
  in the sub-group: Absence of cognitive impairment
Change in spatiotemporal gait, and in particular in the variability of stride time between the two devices | baseline
  in the sub-group: Minor Neurocognitive Disorder
Change in spatiotemporal gait, and in particular in the variability of stride time between the two devices | baseline
  in the sub-group: Major Neurocognitive Disorder

CONTACTS AND LOCATIONS:
Locations (1):
- Angers University Hospital, Angers, France

REFERENCES:
- [Derived] Sacco G, Ben-Sadoun G, Gautier J, Simon R, Goupil M, Laureau P, Terrien J, Annweiler C. Comparison of spatio-temporal gait parameters between the GAITRite(R) platinum plus classic and the GAITRite(R) CIRFACE among older adults: a retrospective observational study. BMC Geriatr. 2023 Mar 7;23(1):132. doi: 10.1186/s12877-023-03811-7. PMID 36882705